CLINICAL TRIAL: NCT01740427
Title: A RANDOMIZED, MULTICENTER, DOUBLE-BLIND PHASE 3 STUDY OF PD-0332991 (ORAL CDK 4/6 INHIBITOR) PLUS LETROZOLE VERSUS PLACEBO PLUS LETROZOLE FOR THE TREATMENT OF POSTMENOPAUSAL WOMEN WITH ER (+), HER2 (-) BREAST CANCER WHO HAVE NOT RECEIVED ANY PRIOR SYSTEMIC ANTI CANCER TREATMENT FOR ADVANCED DISEASE
Brief Title: A Study of Palbociclib (PD-0332991) + Letrozole vs. Letrozole For 1st Line Treatment Of Postmenopausal Women With ER+/HER2- Advanced Breast Cancer (PALOMA-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5481008; 2012-004601-27 (EudraCT Number); PALMOA-2 (Other: Alias Study Number); PALOMA-2 (Other: Alias Study Number)
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; postmenopausal women; estrogen-receptor positive; HER2 negative; locoregionally recurrent; metastatic; Palbociclib (PD-0332991); PALOMA-2
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PD-0332991 + Letrozole (Experimental): PD-0332991, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment in combination with Letrozole, 2.5mg, orally once daily (continuously).
  Interventions: Drug: PD-0332991; Drug: Letrozole
- Placebo + Letrozole (Active Comparator): Placebo, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment in combination with Letrozole, 2.5mg, orally once daily (continuously).
  Interventions: Drug: Placebo; Drug: Letrozole

INTERVENTIONS:
Drug: PD-0332991 — PD-0332991, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Arms: PD-0332991 + Letrozole
Drug: Letrozole — Letrozole, 2.5mg, orally once daily (continuously)
  Arms: PD-0332991 + Letrozole
Drug: Placebo — Placebo, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Arms: Placebo + Letrozole
Drug: Letrozole — Letrozole, 2.5mg, orally once daily (continuously)
  Arms: Placebo + Letrozole

SUMMARY:
The study is designed to compare the clinical benefit following treatment with letrozole in combination with PD-0332991 versus letrozole in combination with placebo in postmenopausal women with ER(+)/HER2(-) advanced breast cancer who have not received prior systemic anti cancer therapies for their advanced/metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with locoregionally recurrent or metastatic disease not amenable to curative therapy.
* Confirmed diagnosis of ER positive breast cancer
* No prior systemic anti-cancer therapy for advanced ER+ disease.
* Postmenopausal women
* Measurable disease as per Response Evaluation Criterion in Solid Tumors [RECIST] or bone-only disease
* Eastern Cooperative Oncology Group [ECOG] 0-2
* Adequate organ and marrow function
* Patient must agree to provide tumor tissue

Exclusion Criteria:

* Confirmed diagnosis of HER2 positive disease
* Patients with advanced, symptomatic, visceral spread that are at risk of life threatening complication in the short term
* Known uncontrolled or symptomatic CNS metastases
* Prior (neo)adjuvant treatment with letrozole or anastrozole with DFI ≤ 12-months from completion of treatment.
* Prior treatment with any CDK 4/6 inhibitor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 666 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2016-02-26 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (299):
- United States (131):
  - Southern California Permanente Medical Group, Bellflower, California
  - Beverly Hills Cancer Center, Beverly Hills, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Los Angeles Hematology/Oncology Medical Group, Glendale, California
  - UCLA Hematology/ Oncology- Irvine, Irvine, California
  - UCLA Hematology Oncology- Laguna Hills, Laguna Hills, California
  - Los Angeles Hematology/Oncology Medical Group, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Translational Research Management, Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy, Attn: Steven L Wong, Pharm.D., Los Angeles, California
  - UCLA West Medical Pharmacy, Attn: Steven L. Wong, Los Angeles, California
  - UCLA West Medical Pharmacy: Drug Management Only, Los Angeles, California
  - UCLA West Medical Pharmacy; Drug Management Only, Los Angeles, California
  - UCLA West Medical Pharmacy, Los Angeles, California
  - Administrative Address: UCLA Hematology/Oncology, Los Angeles, California
  - Drug Management Only: TRIO-US Pharmacy UCLA Medical Plaza, Attn: Steven L Wong, Pharm.D., Los Angeles, California
  - Regulatory Management Only: TRIO-US Central Administration, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - TRIO-US Central Administration: Regulatory Management Only, Los Angeles, California
  - TRIO-US Central Administration, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/ Oncology- Pasadena, Pasadena, California
  - Torrance Health Association, DBa Torrance Memorial Physician Network, Redondo Beach, California
  - Southern California Permanente Medical Group, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of California San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - San Luis Obispo Oncology and Hematology Health Center/ Pacific Central Coast Health Centers, San Luis Obispo, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Santa Monica Medical Center and Orthopaedic Hospital, Santa Monica, California
  - Stanford Women's Cancer Center, Stanford, California
  - Wellness Oncology & Hematology, West Hills, California
  - UCLA Hematology/Oncology- Westlake, Westlake Village, California
  - St. Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Whittingham Cancer Center @ Norwalk Hospital, Norwalk, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sylvester at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Breast Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Cancer Specialist of North Florida, Pharmacy, Jacksonville, Florida
  - Cancer Specialists of North Florida-Southpoint, Jacksonville, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Memorial Breast Cancer Center at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sylvester Comprehensive Cancer Center Plantation, Plantation, Florida
  - Cancer Specialists of North Florida - St. Augustine, Saint Augustine, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Kootenai Clinic Cancer Services, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services, Post Falls, Idaho
  - The Mark M. Connolly Center for Cancer and Specialty Care, Chicago, Illinois
  - Carle Foundation Hospital DBA Carle Cancer Center, Danville, Illinois
  - Carle Foundation Hospital DBA Carle Cancer Center, Effingham, Illinois
  - Presence Infusion Care- Evanston, Evanston, Illinois
  - Carle Foundation Hospital DBA Carle Cancer Center, Mattoon, Illinois
  - Presence Infusion Care- Skokie, Skokie, Illinois
  - Carle Foundation Hospital DBA Carle Cancer Center, Urbana, Illinois
  - James Graham Brown Cancer Center and University Hospital, Louisville, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - The West Clinic, PC, Corinth, Mississippi
  - The West Clinic, PC dba West Cancer Centre, Southaven, Mississippi
  - Mercy Clinic St. Louis Cancer and Breast Institute, Ballwin, Missouri
  - Mercy Clinic St. Louis Cancer and Breast Institute, St Louis, Missouri
  - Mercy Hospital St. Louis - David C. Pratt Cancer Center, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Saint Francis Medical Center, Grand Island, Nebraska
  - Saint Francis Medical Center, Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Saint Francis Medical Center, Hastings, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Regulatory Office: Comprehensive Cancer Centers of Nevada Research Department, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - CareMount Medical, Brewster, New York
  - CareMount Medical, Mount Kisco, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University- Cancer Center, Stony Brook, New York
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - OHSU Center for Health and Healing 2, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - OHSU Research Pharmacy Services, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - The West Clinic, PC dba West Cancer Centre, Germantown, Tennessee
  - Tennessee Oncology PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - The West Clinic, PC dba West Cancer Centre, Memphis, Tennessee
  - Tennessee Oncology PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology PLLC, Smyrna, Tennessee
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas oncology-west Texas, El Paso, Texas
  - Texas oncology-West Texas, El Paso, Texas
  - Texas Oncology-west Texas, El Paso, Texas
  - Investigational Products Center (IPC), Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Department of Breast Medical Oncology, Houston, Texas
  - The University of Texas MD Anderson Cancer Center., Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Products Center, Irving, Texas
  - Oncology & Hematology Associates of Southwest Virginia, INC., D.B.A. Blue Rigde Cancer Care, Blacksburg, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Low Moor, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Salem, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, INC., D.B.A. Blue Rigde Cancer Care, Wytheville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Northwest Cancer Specialists P.C., Vancouver, Washington
  - WVU Medicine, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Australia (16):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Laverty Pathology, Port Macquarie, New South Wales
  - Mid North Coast Diagnostic Imaging, Port Macquarie, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Icon Cancer Care, Auchenflower, Queensland
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Icon Cancer Care Corporate Office, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Bendigo Health Care Group, The Bendigo Hospital Campus, Bendigo, Victoria
  - Northern Hospital, Epping, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (8):
  - Gasthuis Zusters Antwerpen - Campus Sint- Augustinus, Wilrijk, Antwerpen
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - Oncologie, Brussels
  - Grand Hopital de Charleroi / Service d'Hematologie et Oncologie, Charleroi
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - CHU Start Tilman, Liège
  - CHR East Belgium - Verviers, Verviers
- Canada (14):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency-Fraser Valley Centre, Surrey, British Columbia
  - British Columbia Cancer Agency-Vancouver Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre, Victoria General Site, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Southlake Regional Health Centre- Stronach Regional Cancer Centre, Newmarket, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - St. Michaels Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre (MUHC), Glen Site, Cedars Cancer Centre, Montreal, Quebec
  - Hopital du Sacre-Coeur, Montreal, Quebec
  - Center Hospitalier Affilie Universitaire de Quebec, Universite Laval, Hopital du Saint Sacrement, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Fakultni nemocnice Hradec Kralove, Klinika onkologie a radiologie, Hradec Králové, Czechia
- France (12):
  - Institut de Cancerologie de l'Ouest- Paul Papin, Anger Cedex 02
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Centre Val d'Aurelle,, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Departement d'Oncologie Medicale, Paris
  - Centre Eugene Marquis, Rennes
  - Hopital Rene Huguenin/Institut Curie, Saint-Cloud
  - Institut de Cancérologie de l'Ouest-Rene Gauducheau, Saint-Herblain
  - Institut Claudius Regaud- Cancer Comprehensive Center- IUCT-O-Medical Oncology Department, Toulouse Cedex-9
  - Institut Gustave Roussy, Villejuif
- Germany (12):
  - IOZ- Munchen, PGM- Studien GmbH, Munich, Bavaria
  - Klinikverbund Sudwest - Kliniken Sidelfingen-Boblingen, Böblingen
  - University Hospital Carl Gustav Carus - Department for Obstetrics and Gynecology., Dresden
  - Universitatsklinikum Erlangen, Frauenklinik, Erlangen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitatsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Gynakologie und Geburtshilfe, Kiel
  - Universitaetsklinikum Magdeburg AOR Universitaetsfrauenklinik, Magdeburg
  - Katholisches Klinikum Mainz, Mainz
  - Rotkreuzklinikum Munchen, Frauenklinik,, Munich
  - Breast Cancer, University of Munich, Grosshadern Hospital, Munich
  - Frauenklinik und Poliklinik Klinikum rechts der Isar, Technische Universitaet Muenchen, München
  - Klinikum Mutterhaus, Trier
- Hungary (11):
  - Szent Margit Korhaz, Budapest
  - Affidea Diagnosztika Kft., Budapest
  - Orszagos Onkologiai Intezet ,, Budapest
  - Országos Onkológiai Intézet "B" Belgyogyaszati osztaly, Budapest
  - Országos Onkológiai Intézet, Nuklearis Medicina Osztaly, Budapest
  - Országos Onkológiai Intézet, Radiologiai Diagnosztikai Osztily, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Onkoradiologiai Osztaly, Győr
  - Josa Andras Teaching Hospital,, Nyíregyháza
  - Szegedi Tudomanyegyetem Altalanos Orvosi Kar, Patologia Intezet, Szeged
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Altalanos Orvostudomanyi Kar, Szeged
  - Diagnoscan Magyarorszag Kft., Szeged
- Ireland (8):
  - Bon Secours Hospital, Cork
  - St. James Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St Vincents University Hospital, Dublin
  - Department of Medical Oncology, Galway
  - Mid Western Regional Hospital, Limerick
  - Waterford Regional Hospital, Waterford
- Italy (7):
  - Azienda Ospedaliero-Universitaria di Bologna, Policlinico Sant'Orsola-Malpighi, Bologna, BO
  - Irccs Irst, Meldola, FC
  - IRCCS - Istituto Europeo di Oncologia, Milan, Milan
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Istituti Fisioterapici Ospitalieri, Roma
  - Ospedale SS Trinita, Sora (FR)
- Japan (15):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kumamoto City Hospital, Kumamoto, Kumamoto
  - Saitama Cancer Center, Kita-adachi-gun, Saitama
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Niigata Cancer Center Hospital 2-15-3, Niigata
  - Iwate Medical University Hospital, Numakunai
  - National Hospital Organization Osaka National Hospital, Osaka
- Poland (3):
  - Europejskie Centrum Zdrowia Otwock, Otwock, Masovian Voivodeship
  - Oncology and Radiotherapy Clinic, Gdansk
  - Niepubliczny Zakład Opieki Zdrowotnej "Onko-Dent" SP.P. G.L. Słomian, Żory
- Russia (12):
  - Regional Budgetary Healthcare Institution Kursk Regional Clinical, Kursk, Kursk Oblast
  - State Budget Healthcate Institution "Leningrad Region Oncology Dispensary", Kuzmolovo, Leningradskaya Oblast'
  - GUZ Republic Clinical Oncology Dispensary of Ministry of Health of Republic of Tatarstan, Kazan'
  - Federal State Budget Institution, Moscow
  - State Budget Healthcare Institution Moscow City Oncology Hospital, Moscow Area
  - Budget Institution of Healthcare, Omsk
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - Non-State Health Care agency "Road Clinical Hospital of PLC" Russian Railways, Saint Petersburg
  - Saint-Petersburg State Budget Healthcare Institution (SBHCI), Saint Petersburg
  - Republican Clinical Hospital n.a. G.G. Kuvatov, Ufa
  - State Budget Medical Institution Republican Clinical Oncology, Ufa
  - SBHI of Republic of Bashkortostan Emergency Hospital, Ufa
- South Korea (6):
  - National Cancer Center, Center for Breast Cancer, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seodaemun-gu, Seoul
  - Seoul National University Hospital / Department of Internal Medicine, Seoul
  - Asan Medical Center, Division of Oncology, Department of Internal Medicine, Seoul
  - Samsung Medical Center, Division of Hematology-Oncology, Department of Medicine, Seoul
- Spain (22):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Fundacion de Alcorcon, Alcorcón, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital de Donostia, Donostia / San Sebastian
  - Complejo Hospitalario de Jaen, Jaén
  - Instituto Catalan de Oncologia L'Hospitalet, L'Hospitalet de Llobregat (Barcelona)
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Centro Oncologico MD Anderson Internacional España, Madrid
  - Hospital Clinico San Carlos, Madrid
  - HOSPITAL Universitario 12 DE OCTUBRE, Madrid
  - Hospital Madrid Universitario Sanchinarro, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano de Oncologia, Valencia
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Mackay Memory Hospital, Taipei
  - Veterans General Hospital-Taipei, Taipei
- Ukraine (10):
  - MI "Dnipropetrovsk City Multidisciplinary Clinical Hospital No.4" of the Dnipropetrovsk City Council, Dnipro
  - State Institution Dnipropetrovsk Medical Academy at the Ministry of Health of Ukraine, Dnipro
  - Municipal Non-profit Enterprise "Regional Centre of Oncology", Kharkiv
  - Lviv State Oncologic Regional Treatment and Diagnostic Center, Chemotherapy Department, Lviv
  - Municipal Medical Institution "Makiivka City Hospital No.2 of Donetsk Region", Makiivka
  - Regional Municipal Establishment "Sumy Regional Clinical Oncology Dispensary", Thoracic Department, Sumy
  - City Oncology Centre of Central Municipal Clinical Hospital, Uzhhorod
  - Institute of Postgraduate education and preuniversity preparing of Uzhgorod National Univ., Uzhhorod
  - MI "Zaporizhzhia Regional Clinical Oncology Dispensary" Zaporizhzhia Regional Assembly,, Zaporizhzhia
  - State institution "Zaporizhzhia Medical Academy of Postgraduate Education MOH Ukraine",, Zaporizhzhya
- United Kingdom (8):
  - Kent Oncology Center, Maidstone, KENT
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh, Scotland
  - Beatson Institute for Cancer Research, Glasgow, Scotland
  - Guys Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - Charing Cross Hospital, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - The Research And Development Office, The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cheang MCU, Rimawi M, Johnston S, Jacobs SA, Bliss J, Pogue-Geile K, Kilburn L, Zhu Z, Schuster EF, Xiao H, Swaim L, Deng S, Lu DR, Gauthier E, Tursi J, Slamon DJ, Rugo HS, Finn RS, Liu Y. Effect of cross-platform gene-expression, computational methods on breast cancer subtyping in PALOMA-2 and PALLET studies. NPJ Breast Cancer. 2024 Jun 29;10(1):54. doi: 10.1038/s41523-024-00658-y. PMID 38951507
- [Derived] Li H, Wu Y, Zou H, Koner S, Plichta JK, Tolaney SM, Zhang J, He YW, Wei Q, Tang L, Zhang H, Zhang B, Guo Y, Chen X, Li K, Lian L, Ma F, Luo S. Clinical efficacy of CDK4/6 inhibitor plus endocrine therapy in HR-positive/HER2-0 and HER2-low-positive metastatic breast cancer: a secondary analysis of PALOMA-2 and PALOMA-3 trials. EBioMedicine. 2024 Jul;105:105186. doi: 10.1016/j.ebiom.2024.105186. Epub 2024 Jun 10. PMID 38861871
- [Derived] Slamon DJ, Dieras V, Rugo HS, Harbeck N, Im SA, Gelmon KA, Lipatov ON, Walshe JM, Martin M, Chavez-MacGregor M, Bananis E, Gauthier E, Lu DR, Kim S, Finn RS. Overall Survival With Palbociclib Plus Letrozole in Advanced Breast Cancer. J Clin Oncol. 2024 Mar 20;42(9):994-1000. doi: 10.1200/JCO.23.00137. Epub 2024 Jan 22. PMID 38252901
- [Derived] Jhaveri K, O'Shaughnessy J, Fasching PA, Tolaney SM, Yardley DA, Sharma VK, Biswas C, Thuerigen A, Pathak P, Rugo HS. Matching-adjusted indirect comparison of PFS and OS comparing ribociclib plus letrozole versus palbociclib plus letrozole as first-line treatment of HR+/HER2- advanced breast cancer. Ther Adv Med Oncol. 2023 Dec 14;15:17588359231216095. doi: 10.1177/17588359231216095. eCollection 2023. PMID 38107828
- [Derived] Rugo HS, Im SA, Joy AA, Shparyk Y, Walshe JM, Sleckman B, Loi S, Theall KP, Kim S, Huang X, Bananis E, Mahtani R, Finn RS, Dieras V. Effect of palbociclib plus endocrine therapy on time to chemotherapy across subgroups of patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: Post hoc analyses from PALOMA-2 and PALOMA-3. Breast. 2022 Dec;66:324-331. doi: 10.1016/j.breast.2022.11.005. Epub 2022 Nov 15. PMID 36463643
- [Derived] Zhu Z, Turner NC, Loi S, Andre F, Martin M, Dieras V, Gelmon KA, Harbeck N, Zhang C, Cao JQ, Yan Z, Lu DR, Wei P, VanArsdale TL, Rejto PA, Huang X, Rugo HS, Loibl S, Cristofanilli M, Finn RS, Liu Y. Comparative biomarker analysis of PALOMA-2/3 trials for palbociclib. NPJ Precis Oncol. 2022 Aug 16;6(1):56. doi: 10.1038/s41698-022-00297-1. PMID 35974168
- [Derived] Gelmon K, Walshe JM, Mahtani R, Joy AA, Karuturi M, Neven P, Lu DR, Kim S, Schnell P, Bananis E, Schwartzberg L. Efficacy and safety of palbociclib in patients with estrogen receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer with preexisting conditions: A post hoc analysis of PALOMA-2. Breast. 2021 Oct;59:321-326. doi: 10.1016/j.breast.2021.07.017. Epub 2021 Jul 28. PMID 34388698
- [Derived] Iwata H, Umeyama Y, Liu Y, Zhang Z, Schnell P, Mori Y, Fletcher O, Marshall JC, Johnson JG, Wood LS, Toi M, Finn RS, Turner NC, Bartlett CH, Cristofanilli M. Evaluation of the Association of Polymorphisms With Palbociclib-Induced Neutropenia: Pharmacogenetic Analysis of PALOMA-2/-3. Oncologist. 2021 Jul;26(7):e1143-e1155. doi: 10.1002/onco.13811. Epub 2021 Jun 7. PMID 33955129
- [Derived] Finn RS, Rugo HS, Gelmon KA, Cristofanilli M, Colleoni M, Loi S, Schnell P, Lu DR, Theall KP, Mori A, Gauthier E, Bananis E, Turner NC, Dieras V. Long-Term Pooled Safety Analysis of Palbociclib in Combination with Endocrine Therapy for Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Updated Analysis with up to 5 Years of Follow-Up. Oncologist. 2021 May;26(5):e749-e755. doi: 10.1002/onco.13684. Epub 2021 Mar 10. PMID 33486783
- [Derived] Zheng J, Yu Y, Durairaj C, Dieras V, Finn RS, Wang DD. Impact of Dose Reduction on Efficacy: Implications of Exposure-Response Analysis of Palbociclib. Target Oncol. 2021 Jan;16(1):69-76. doi: 10.1007/s11523-020-00771-5. PMID 33211314
- [Derived] Finn RS, Cristofanilli M, Ettl J, Gelmon KA, Colleoni M, Giorgetti C, Gauthier E, Liu Y, Lu DR, Zhang Z, Bartlett CH, Slamon DJ, Turner NC, Rugo HS. Treatment effect of palbociclib plus endocrine therapy by prognostic and intrinsic subtype and biomarker analysis in patients with bone-only disease: a joint analysis of PALOMA-2 and PALOMA-3 clinical trials. Breast Cancer Res Treat. 2020 Nov;184(1):23-35. doi: 10.1007/s10549-020-05782-4. Epub 2020 Aug 11. PMID 32783178
- [Derived] Huang Bartlett C, Mardekian J, Cotter MJ, Huang X, Zhang Z, Parrinello CM, Bourla AB. Concordance of real-world versus conventional progression-free survival from a phase 3 trial of endocrine therapy as first-line treatment for metastatic breast cancer. PLoS One. 2020 Apr 21;15(4):e0227256. doi: 10.1371/journal.pone.0227256. eCollection 2020. PMID 32315295
- [Derived] Ettl J, Im SA, Ro J, Masuda N, Colleoni M, Schnell P, Bananis E, Lu DR, Cristofanilli M, Rugo HS, Finn RS. Hematologic adverse events following palbociclib dose reduction in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: pooled analysis from randomized phase 2 and 3 studies. Breast Cancer Res. 2020 Mar 12;22(1):27. doi: 10.1186/s13058-020-01263-0. PMID 32164785
- [Derived] Rugo HS, Finn RS, Gelmon K, Joy AA, Harbeck N, Castrellon A, Mukai H, Walshe JM, Mori A, Gauthier E, Lu DR, Bananis E, Martin M, Dieras V. Progression-free Survival Outcome Is Independent of Objective Response in Patients With Estrogen Receptor-positive, Human Epidermal Growth Factor Receptor 2-negative Advanced Breast Cancer Treated With Palbociclib Plus Letrozole Compared With Letrozole: Analysis From PALOMA-2. Clin Breast Cancer. 2020 Apr;20(2):e173-e180. doi: 10.1016/j.clbc.2019.08.009. Epub 2019 Sep 5. PMID 31836434
- [Derived] Dieras V, Harbeck N, Joy AA, Gelmon K, Ettl J, Verma S, Lu DR, Gauthier E, Schnell P, Mori A, Rugo HS, Finn RS. Palbociclib with Letrozole in Postmenopausal Women with ER+/HER2- Advanced Breast Cancer: Hematologic Safety Analysis of the Randomized PALOMA-2 Trial. Oncologist. 2019 Dec;24(12):1514-1525. doi: 10.1634/theoncologist.2019-0019. Epub 2019 Jun 19. PMID 31217344
- [Derived] Masuda N, Mukai H, Inoue K, Rai Y, Ohno S, Mori Y, Hashigaki S, Muramatsu Y, Umeyama Y, Iwata H, Toi M. Neutropenia management with palbociclib in Japanese patients with advanced breast cancer. Breast Cancer. 2019 Sep;26(5):637-650. doi: 10.1007/s12282-019-00970-7. Epub 2019 May 24. PMID 31127500
- [Derived] Im SA, Mukai H, Park IH, Masuda N, Shimizu C, Kim SB, Im YH, Ohtani S, Huang Bartlett C, Lu DR, Iyer S, Mori Y, Mori A, Gauthier E, Finn RS, Toi M. Palbociclib Plus Letrozole as First-Line Therapy in Postmenopausal Asian Women With Metastatic Breast Cancer: Results From the Phase III, Randomized PALOMA-2 Study. J Glob Oncol. 2019 May;5:1-19. doi: 10.1200/JGO.18.00173. PMID 31125276
- [Derived] Rugo HS, Finn RS, Dieras V, Ettl J, Lipatov O, Joy AA, Harbeck N, Castrellon A, Iyer S, Lu DR, Mori A, Gauthier ER, Bartlett CH, Gelmon KA, Slamon DJ. Palbociclib plus letrozole as first-line therapy in estrogen receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer with extended follow-up. Breast Cancer Res Treat. 2019 Apr;174(3):719-729. doi: 10.1007/s10549-018-05125-4. Epub 2019 Jan 10. PMID 30632023
- [Derived] Mukai H, Shimizu C, Masuda N, Ohtani S, Ohno S, Takahashi M, Yamamoto Y, Nishimura R, Sato N, Ohsumi S, Iwata H, Mori Y, Hashigaki S, Muramatsu Y, Nagasawa T, Umeyama Y, Lu DR, Toi M. Palbociclib in combination with letrozole in patients with estrogen receptor-positive, human epidermal growth factor receptor 2-negative advanced breast cancer: PALOMA-2 subgroup analysis of Japanese patients. Int J Clin Oncol. 2019 Mar;24(3):274-287. doi: 10.1007/s10147-018-1353-9. Epub 2018 Dec 4. PMID 30515674
- [Derived] Rugo HS, Turner NC, Finn RS, Joy AA, Verma S, Harbeck N, Masuda N, Im SA, Huang X, Kim S, Sun W, Iyer S, Schnell P, Bartlett CH, Johnston S. Palbociclib plus endocrine therapy in older women with HR+/HER2- advanced breast cancer: a pooled analysis of randomised PALOMA clinical studies. Eur J Cancer. 2018 Sep;101:123-133. doi: 10.1016/j.ejca.2018.05.017. Epub 2018 Jul 25. PMID 30053671
- [Derived] Dieras V, Rugo HS, Schnell P, Gelmon K, Cristofanilli M, Loi S, Colleoni M, Lu DR, Mori A, Gauthier E, Huang Bartlett C, Slamon DJ, Turner NC, Finn RS. Long-term Pooled Safety Analysis of Palbociclib in Combination With Endocrine Therapy for HR+/HER2- Advanced Breast Cancer. J Natl Cancer Inst. 2019 Apr 1;111(4):419-430. doi: 10.1093/jnci/djy109. PMID 30032196
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361
- [Derived] Rugo HS, Dieras V, Gelmon KA, Finn RS, Slamon DJ, Martin M, Neven P, Shparyk Y, Mori A, Lu DR, Bhattacharyya H, Bartlett CHUANG, Iyer S, Johnston S, Ettl J, Harbeck N. Impact of palbociclib plus letrozole on patient-reported health-related quality of life: results from the PALOMA-2 trial. Ann Oncol. 2018 Apr 1;29(4):888-894. doi: 10.1093/annonc/mdy012. PMID 29360932
- [Derived] Turner NC, Finn RS, Martin M, Im SA, DeMichele A, Ettl J, Dieras V, Moulder S, Lipatov O, Colleoni M, Cristofanilli M, Lu DR, Mori A, Giorgetti C, Iyer S, Bartlett CH, Gelmon KA. Clinical considerations of the role of palbociclib in the management of advanced breast cancer patients with and without visceral metastases. Ann Oncol. 2018 Mar 1;29(3):669-680. doi: 10.1093/annonc/mdx797. PMID 29342248
- [Derived] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- See also: To obtain contact information for a study center near you, click here. — https://www.pmiform.com/clinical-trial-info-request?StudyID=A5481008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 666 participants were randomized at 239 centers in 19 countries.
Pre-assignment Details: The study consisted of a screening visit within 28 days before randomization, an active treatment phase, divided in cycles of 28 days each, and a post-treatment follow-up period during which survival and new anti-cancer therapy information was collected every 6 months (±7 days) from the last dose of study treatment.
Groups:
- Palbociclib Plus Letrozole: Participants received letrozole 2.5 milligram (mg) orally QD (once daily) combined with palbociclib 125 mg QD for 21 days of every-28-day cycle, followed by 7 days off treatment.
- Placebo Plus Letrozole: Participants received letrozole 2.5 mg orally QD combined with placebo QD for 21 days of every-28-day cycle, followed by 7 days off treatment.
Period: Overall Study
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Started | 444 | 222
Completed | 0 | 0
Not Completed | 444 | 222
Not completed — Objective Progression or Relapse | 286 | 172
Not completed — Adverse Event | 32 | 9
Not completed — Global Deterioration of Health Status | 28 | 12
Not completed — Participant Refused Continued Treatment | 27 | 15
Not completed — Unspecified reasons | 52 | 8
Not completed — Death | 10 | 3
Not completed — Protocol Violation | 5 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Site Terminated by Sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole | Total
Number analyzed (Participants) | 444 | 222 | 666
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (10.6) | 60.6 (11.2) | 61.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 444 | 222 | 666
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator
Description: PFS is defined as the time from the date of randomization to the date of the first documentation of objective tumor progression as per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) or death due to any cause in the absence of documented PD, whichever occurs first. If tumor progression data include more than 1 date, the first date will be used. PFS (in months) will be calculated as (first event date - randomization date +1)/30.4. Progression is defined using RECIST v1.1, as a 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions, or the appearance of new lesions.
Time Frame: From randomization date to date of first documentation of progression or death (up to approximately 2.5 years)
Population: ITT population or full analysis set included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study medication or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Months | 24.8 [22.1 to NA] — The value was not available because there was not enough disease progression events in the treatment group at the time of analysis, due to drug benefit. | 14.5 [12.9 to 17.1]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Test type: Superiority or Other; p < 0.000001, Stratified Log Rank — 1-sided p-value from the stratified log-rank test; Hazard Ratio (HR) = 0.576, 95% CI 2-sided [0.463 to 0.718]

2. Secondary Outcome: Objective Response as Assessed by the Investigator
Description: Objective Response (OR) defined as overall complete response (CR) or partial response (PR) according to RECIST v1.1. Objective Response Rate (ORR) is defined as proportion of participants with CR or PR relative to all randomized participants with measurable disease at baseline. Participants who do not have on-study radiographic tumor re-evaluation, who received anti-tumor treatment, or who died, progressed/ dropped out for any reason prior to reaching a CR or PR were counted as non-responders in assessment of ORR. Per RECIST v1.1, CR: Complete disappearance of target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10mm). PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter is used in the sum for target nodes, while the longest diameter is used in the sum for all other target lesions. Stable Disease: neither sufficient shrinkage nor increase to qualify for disease progression.
Time Frame: From randomization until end of treatment (up to approximately 2.5 years)
Population: ITT population or full analysis set included all participants who were randomized, with study medication, regardless of whether participants received study medication or received a different drug from that to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Percentage of participants | 46.4 [41.7 to 51.2] | 38.3 [31.9 to 45.0]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Stratified analysis: Stratified by disease site (visceral vs non-visceral) per randomization; Test type: Superiority or Other; p = 0.0224, Fisher Exact — 1-sided p-value is from exact test; Odds Ratio (OR) = 1.428, 95% CI 2-sided [1.008 to 2.030]

3. Secondary Outcome: Objective Response: Participants With Measurable Disease at Baseline as Assessed by the Investigator
Description: The OR is defined as the overall CR or PR according to the RECIST v1.1. ORR is defined as proportion of participants with CR or PR relative to all randomized participants with measurable disease at baseline. Participants who do not have on-study radiographic tumor re-evaluation, who received anti-tumor treatment, or who died, progressed/ dropped out for any reason prior to reaching a CR or PR were counted as non-responders in the assessment of ORR. Per RECIST v1.1, CR: Complete disappearance of target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10mm). PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter is used in the sum for target nodes, while the longest diameter is used in the sum for all other target lesions. Stable Disease: neither sufficient shrinkage nor increase to qualify for disease progression.
Time Frame: From randomization until end of treatment (up to approximately 2.5 years)
Population: Participants who had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 338 | 171
Percentage of participants | 60.7 [55.2 to 65.9] | 49.1 [41.4 to 56.9]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Stratified analysis: Stratified by disease site (visceral vs non-visceral) per randomization; Test type: Superiority or Other; p = 0.0090, Fisher Exact — 1-sided p-value is from exact test; Odds Ratio (OR) = 1.594, 95% CI 2-sided [1.080 to 2.347]

4. Secondary Outcome: Duration of Response (DR)
Description: DR is defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurs first. If tumor progression data included more than 1 date, the first date will be used. DR was calculated as [the date response ended (i.e. date of PD or death) - first CR or PR date + 1)]/30.4. DR would only be calculated for the subgroup of participants with an objective tumor response. Per RECIST v1.1, CR: Complete disappearance of target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10mm). PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions.The short diameter is used in the sum for target nodes, while the longest diameter is used in the sum for all other target lesions. Stable Disease: neither sufficient shrinkage nor increase to qualify for disease progression.
Time Frame: From randomization until end of treatment (up to approximately 2.5 years)
Population: Participants who had tumor response with CR or PR during study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 206 | 85
Months | 20.1 [19.3 to 28.0] | 16.7 [13.8 to 22.5]

5. Secondary Outcome: Disease Control (DC)/Clinical Benefit Response (CBR)
Description: DC is defined as overall CR, PR, or stable disease (SD) >=24 weeks according to RECIST version 1.1. Disease Control Rate (DCR) is defined as participants with CR, PR, or SD >=24 weeks relative to all randomized participants. Participants who do not have on-study radiographic tumor reevaluation, who received anti-tumor treatment, a best response of SD>=24 weeks, or who died, progressed, or dropped out for any reason prior to achieving reaching a CR or PR and a best response of SD>=24 weeks was counted as non-responders in DCR. Per RECIST v1.1, CR: Complete disappearance of target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10mm). PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter is used in the sum for target nodes, while the longest diameter is used in the sum for all other target lesions. SD: neither sufficient shrinkage nor increase to qualify for disease progression.
Time Frame: From randomization until end of treatment (up to approximately 2.5 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Percentage of participants | 85.8 [82.2 to 88.9] | 71.2 [64.7 to 77.0]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Stratified analysis: Stratified by disease site (visceral, non-visceral) per randomization; Test type: Superiority or Other; p < 0.0001, Fisher Exact — 1-sided p-value is from exact test; Odds Ratio (OR) = 2.451, 95% CI 2-sided [1.619 to 3.722]

6. Secondary Outcome: PFS by Tumor Tissue Biomarkers Status, Including Genes (eg, Copy Numbers of CCND1, CDKN2A), Proteins (eg, Ki67, pRb), and RNA Expression (eg, cdk4, cdk6)
Description: PFS by biomarker status by Investigator assessment. Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Positive is defined as H-Score >=1 and negative as H-Score <1. H-Score is calculated as the sum of the % of cells at each level of staining intensity (0, 1+, 2+, and 3+) multiplied by the staining intensity value: H-Score = (% at 0)*0 + (% at 1+)*1 + (% at 2+)*2 + (% at 3+)*3. H-Score values range from 0 to 300. ER stands for estrogen receptor and Rb stands for retinoblastoma susceptibility gene product.
Time Frame: From randomization until end of treatment (up to approximately 24 Months)
Population: ITT population or full analysis set included all participants who were randomized, with study medication, regardless of whether participants received study medication or received a different drug from that to which they were randomized. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Months
  ER Positive: number analyzed (Participants) | 338 | 166
  ER Positive | 24.9 [22.2 to NA] — Not reached; insufficient number of participants with events. | 16.3 [12.9 to 19.1]
  ER Negative: number analyzed (Participants) | 40 | 22
  ER Negative | 15.6 [8.3 to 22.0] | 5.4 [2.7 to 11.1]
  Rb Positive: number analyzed (Participants) | 345 | 167
  Rb Positive | 24.2 [21.4 to 25.7] | 13.7 [11.0 to 16.5]
  Rb Negative: number analyzed (Participants) | 29 | 22
  Rb Negative | NA [11.4 to NA] — Not reached; insufficient number of participants with events. | 18.5 [2.9 to NA] — Not reached; insufficient number of participants with events.
  Cyclin D1 Positive: number analyzed (Participants) | 370 | 179
  Cyclin D1 Positive | 24.8 [21.5 to 27.6] | 13.8 [11.3 to 16.8]
  Cyclin D1 Negative: number analyzed (Participants) | 5 | 10
  Cyclin D1 Negative | 11.1 [2.2 to 23.9] | 8.1 [0.4 to NA] — Not reached; insufficient number of participants with events.
  p16 Positive: number analyzed (Participants) | 305 | 161
  p16 Positive | 24.8 [21.5 to NA] — Not reached; insufficient number of participants with events. | 13.8 [11.1 to 16.8]
  p16 Negative: number analyzed (Participants) | 59 | 25
  p16 Negative | 16.8 [11.1 to 24.9] | 13.8 [8.1 to NA] — Not reached; insufficient number of participants with events.
  p16 H-Score<175: number analyzed (Participants) | 341 | 177
  p16 H-Score<175 | 23.7 [19.6 to 25.7] | 13.8 [11.2 to 16.8]
  p16 H-Score>=175: number analyzed (Participants) | 23 | 9
  p16 H-Score>=175 | 24.2 [11.1 to NA] — Not reached; insufficient number of participants with events. | 5.6 [1.5 to 19.1]
  Ki67 <=20%: number analyzed (Participants) | 216 | 102
  Ki67 <=20% | 27.6 [24.2 to NA] — Not reached; insufficient number of participants with events. | 16.8 [13.7 to 22.0]
  Ki67 >20%: number analyzed (Participants) | 152 | 83
  Ki67 >20% | 17.5 [13.8 to 22.0] | 8.4 [5.6 to 13.6]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for ER positive; Test type: Superiority or Other; p < 0.0001, Unstratified log-rank test; Hazard Ratio (HR) = 0.571, 95% CI 2-sided [0.443 to 0.737] — Unstratified Cox proportional hazards model was used
Statistical Analysis 2: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for ER Negative; Test type: Superiority or Other; p = 0.0030, Unstratified log-rank test; Hazard Ratio (HR) = 0.405, 95% CI 2-sided [0.218 to 0.751] — Unstratified Cox proportional hazards model was used
Statistical Analysis 3: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for Rb Positive; Test type: Superiority or Other; p < 0.0001, Unstratified log-rank test; Hazard Ratio (HR) = 0.531, 95% CI 2-sided [0.416 to 0.680] — Unstratified Cox proportional hazards model was used
Statistical Analysis 4: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for Rb Negative; Test type: Superiority or Other; p = 0.3237, Unstratified log-rank test; Hazard Ratio (HR) = 0.675, 95% CI 2-sided [0.308 to 1.481] — Unstratified Cox proportional hazards model was used
Statistical Analysis 5: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for Cyclin D1 Positive; Test type: Superiority or Other; p < 0.0001, Unstratified log-rank test; Hazard Ratio (HR) = 0.555, 95% CI 2-sided [0.437 to 0.705] — Unstratified Cox proportional hazards model was used
Statistical Analysis 6: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for Cyclin D1 Negative; Test type: Superiority or Other; p = 0.9964, Unstratified log-rank test; Hazard Ratio (HR) = 0.997, 95% CI 2-sided [0.287 to 3.461] — Unstratified Cox proportional hazards model was used
Statistical Analysis 7: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for p16 Positive; Test type: Superiority or Other; p < 0.0001, Unstratified log-rank test; Hazard Ratio (HR) = 0.518, 95% CI 2-sided [0.400 to 0.670] — Unstratified Cox proportional hazards model was used
Statistical Analysis 8: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for p16 Negative; Test type: Superiority or Other; p = 0.3221, Unstratified log-rank test; Hazard Ratio (HR) = 0.731, 95% CI 2-sided [0.392 to 1.364] — Unstratified Cox proportional hazards model was used
Statistical Analysis 9: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for p16 HScore<175; Test type: Superiority or Other; p < 0.0001, Unstratified log-rank test; Hazard Ratio (HR) = 0.581, 95% CI 2-sided [0.455 to 0.742] — Unstratified Cox proportional hazards model was used
Statistical Analysis 10: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for p16 HScore>=175; Test type: Superiority or Other; p = 0.0022, Unstratified log-rank test; Hazard Ratio (HR) = 0.255, 95% CI 2-sided [0.100 to 0.650] — Unstratified Cox proportional hazards model was used
Statistical Analysis 11: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for Ki67 <=20%; Test type: Superiority or Other; p = 0.0002, Unstratified log-rank test; Hazard Ratio (HR) = 0.530, 95% CI 2-sided [0.379 to 0.742] — Unstratified Cox proportional hazards model was used
Statistical Analysis 12: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Statistical analysis for Ki67 >20%; Test type: Superiority or Other; p = 0.0007, Unstratified log-rank test; Hazard Ratio (HR) = 0.569, 95% CI 2-sided [0.409 to 0.791] — Unstratified Cox proportional hazards model was used

7. Secondary Outcome: Corrected QT Interval (QTc) Time-Matched Change From Baseline on Cycle 1 Day 14
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and sent to a central laboratory for blinded manual adjudication. The average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR), by Bazette's formula (QTcB = QT divided by square root of RR) and corrected QT interval according to study-specific criteria (QTcS). Time-matched change from baseline values were reported for QTc analysis population.
Time Frame: Time-matched triplicate ECGs were collected at 0 (predose), 2, 4, 6 and 8 hours on Day 0 and on Cycle1 Day14
Population: QTc analysis set is a subset of as treated (AT) population who were in Group 1; their QTc was used to study the effect of palbociclib on QT interval via serial triplicate ECGs with PK draws; and who had >= 1 pair of time-matched Day 0 and palbociclib postdose (Cycle1 Day14) measurements.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 76 | 47
msec
  QTcS at 0 hour | 0.80 [-1.67 to 3.26] | 2.95 [-0.19 to 6.10]
  QTcS at 2 hour | 3.32 [0.79 to 5.85] | 1.65 [-1.48 to 4.78]
  QTcS at 4 hour | 2.76 [0.23 to 5.30] | 1.74 [-1.39 to 4.87]
  QTcS at 6 hour | 4.49 [1.96 to 7.02] | 0.72 [-2.41 to 3.85]
  QTcS at 8 hour | 0.94 [-1.60 to 3.48] | 3.14 [0.01 to 6.27]
  QTcF at 0 hour | 1.10 [-1.39 to 3.58] | 3.06 [-0.11 to 6.23]
  QTcF at 2 hour | 3.68 [1.12 to 6.23] | 1.73 [-1.43 to 4.88]
  QTcF at 4 hour | 2.86 [0.31 to 5.41] | 1.54 [-1.62 to 4.70]
  QTcF at 6 hour | 4.57 [2.01 to 7.12] | 0.71 [-2.44 to 3.87]
  QTcF at 8 hour | 1.21 [-1.36 to 3.77] | 2.84 [-0.31 to 6.00]
  QTcB at 0 hour | -0.11 [-2.83 to 2.61] | 2.78 [-0.69 to 6.25]
  QTcB at 2 hour | 1.46 [-1.34 to 4.25] | 0.83 [-2.63 to 4.28]
  QTcB at 4 hour | 2.58 [-0.22 to 5.38] | 2.47 [-0.98 to 5.92]
  QTcB at 6 hour | 4.03 [1.24 to 6.83] | 0.53 [-2.92 to 3.99]
  QTcB at 8 hour | -0.17 [-2.98 to 2.64] | 4.14 [0.69 to 7.59]

8. Secondary Outcome: Percentage of Participants With Corrected QT Interval (QTc)
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and sent to a central laboratory for blinded manual adjudication. The average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR), by Bazette's formula (QTcB = QT divided by square root of RR) and corrected QT interval according to study-specific criteria (QTcS). Percentage of participants with post-baseline maximum absolute values and maximum increase from baseline were summarized for the safety analysis population.
Time Frame: For safety monitoring triplicate ECGs were obtained at 0 hour (pre-dose) on Day 1 of Cycle 1, Day 14 of Cycles 1 and Cycle 2, then on Day 1 of Cycles 4, 7, and 10 (ECGs beyond Cycle 10 were performed as clinically indicated)
Population: The AT population or safety analysis set included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 441 | 220
Percentage of participants
  Maximum QTcS <450 msec | 80.5 | 85.9
  Maximum QTcS 450-<480 msec | 17.9 | 11.8
  Maximum QTcS 480-<500 msec | 1.1 | 2.3
  Maximum QTcS >=500 msec | 0.5 | 0
  Maximum QTcF <450 msec | 85.9 | 89.5
  Maximum QTcF 450-<480 msec | 12.2 | 9.5
  Maximum QTcF 480-<500 msec | 1.6 | 0.9
  Maximum QTcF >=500 msec | 0.2 | 0
  Maximum QTcB <450 msec | 64.9 | 69.1
  Maximum QTcB 450-<480 msec | 32.2 | 27.3
  Maximum QTcB 480-<500 msec | 2.3 | 3.2
  Maximum QTcB >=500 msec | 0.7 | 0.5
  Maximum QTcS Change <30 msec | 92.7 | 94.5
  Maximum QTcS 30<=Change <60 msec | 6.6 | 5.5
  Maximum QTcS Change>=60 msec | 0.7 | 0
  Maximum QTcF Change <30 msec | 91.6 | 93.6
  Maximum QTcF 30<=Change <60 msec | 7.9 | 6.4
  Maximum QTcF Change>=60 msec | 0.5 | 0
  Maximum QTcB Change <30 msec | 88.9 | 91.4
  Maximum QTcB 30<=Change <60 msec | 10.2 | 8.2
  Maximum QTcB Change>=60 msec | 0.9 | 0.5

9. Secondary Outcome: Observed Plasma Trough Concentration (Ctrough) at Steady-State
Description: Summary of plasma palbociclib within-participant mean steady-state trough concentrations.
Time Frame: 0 hour (predose) on Day 14 of cycles 1 and 2
Population: Pharmacokinetic analysis set was a subset of AT participants, who were treated with Palbociclib and had at least one measured plasma concentration. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Palbociclib Plus Letrozole
Number analyzed (Participants) | 423
Nanogram per milliliter (ng/mL)
  Cycle 1 Day 14: number analyzed (Participants) | 395
  Cycle 1 Day 14 | 70.1 (59)
  Cycle 2 Day 14: number analyzed (Participants) | 401
  Cycle 2 Day 14 | 64.2 (82)

10. Secondary Outcome: Change From Baseline Between Treatment Comparison in Euro Quality of Life (EQ-5D) Index
Description: The EuroQol EQ-5D is a 6-item instrument designed to assess health status in terms of a single index value or utility score. It contains 5 descriptors of current health state (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with each dimension having 3 levels of function (1=no problem, 2=some problem, and 3=extreme problem). The scores on the 5 descriptors are summarized to create a single summary score. An overall utility score is calculated based on these domains, with a range score from 0 (worse health scenario) to a maximum of 1.0 (best health scenario).
Time Frame: From Baseline up to 2.5 years
Population: Patient Reported Outcome (PRO) Analysis Set is a subset of ITT participants, who had both baseline and at least one follow-up PRO assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 437 | 218
Units on a scale | 0.014 [0.00 to 0.03] | -0.010 [-0.03 to 0.01]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Test type: Superiority or Other; p = 0.0925, Mixed Models Analysis; Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.004 to 0.051]

11. Secondary Outcome: Change From Baseline Between Treatment Comparison in Functional Assessment of Cancer Therapy-Breast (FACT-B)
Description: FACT is a modular approach to assess participant health-related quality of life using a 'core' set of questions (FACT-G) as well as a cancer site-specific module. The FACT-G is a 27-item compilation of general questions divided into 4 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. The FACT-B consisted of the FACT-G (27-item) and a breast-specific module: a 10-item instrument designed to assess participant concerns relating to breast cancer. For all questions, participants were asked to respond to a five-level scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much. FACT-B total score = Physical Well-Being + Social/Family Well-Being + Emotional Well-Being + Functional Well-Being + Breast Cancer Subscale. As each of the items ranges from 0-4, the range of possible scores is 0-144, with 0 being the worst possible score and 144 the best.
Time Frame: From Baseline up to 2.5 years
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 439 | 218
Units on a scale | -0.106 [-1.42 to 1.21] | 0.219 [-1.68 to 2.12]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Test type: Superiority or Other; p = 0.7822, Mixed Models Analysis; [statistical method as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.325, 95% CI 2-sided [-2.63 to 1.98]

12. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs): All Causalities
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. SAE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization; resulted in persistent or significant disability or in congenital anomaly/birth defect. TEAE were events that occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Severity was graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0 as Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening and Grade 5 = death related to AE. Discontinuation included permanent, temporary discontinuation and dose reduction due to AEs.
Time Frame: From date of randomization up to 28 days after last dose of study drug (final analysis till study completion, approximately up to 10.51 years)
Population: AT population included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Percentage of participants
  Participants with AEs | 99.1 | 96.4
  Participants with SAEs | 28.2 | 17.1
  Participants with Grade 3 or 4 AEs | 83.1 | 30.2
  Participants with Grade 5 AEs | 3.6 | 2.3
  Permanently discontinued study due to AEs | 4.1 | 2.3
  Permanently disc. palbociclib/placebo due to AEs | 14.4 | 6.3
  Permanently discontinued letrozole due to AEs | 9.2 | 5.9
  Temporarily disc. palbociclib/placebo due to AEs | 79.7 | 17.1
  Temporarily discontinued letrozole due to AEs | 23.0 | 11.3
  With palbociclib/placebo dose reduction due to AEs | 41.9 | 2.3

13. Secondary Outcome: Overall Survival (OS): Primary Analysis
Description: OS was defined as the time from date of randomization to date of death due to any cause. Participants without survival data beyond the date of their last follow-up were censored on the last date they were known to be alive. Data for this outcome measure was reported at primary analysis.
Time Frame: From date of randomization until death due to any cause or censored, (assessed up to data cut-off date of 15-Nov-2021, approximately 8.7 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Months | 53.9 [49.8 to 60.8] | 51.2 [43.7 to 58.9]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Test type: Superiority or Other; p = 0.337750, Stratified Log Rank — 1-sided p-value from the stratified log-rank test; Hazard Ratio (HR) = 0.956, 95% CI 2-sided [0.777 to 1.177]

14. Secondary Outcome: Overall Survival (OS): Final Analysis
Description: OS was defined as the time from date of randomization to date of death due to any cause. Participants without survival data beyond the date of their last follow-up were censored on the last date they were known to be alive. Data for this outcome measure was reported at final analysis.
Time Frame: From date of randomization until death due to any cause or censored (final analysis till study completion, approximately up to 10.51 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Months | 53.8 [49.8 to 59.2] | 49.8 [42.3 to 56.4]
Statistical Analysis 1: Comparison: Palbociclib Plus Letrozole vs Placebo Plus Letrozole; Test type: Superiority or Other; p = 0.208706, Stratified Log Rank — 1-sided p-value from the stratified log-rank test; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.755 to 1.124]

15. Secondary Outcome: Survival Probability at 1 Year, 2 Year and 3 Year
Description: One, two or three-year survival probability was defined as the probability of survival 1 year, 2 or 3 years after the date of randomization. The survival probability was estimated using the Kaplan-Meier method and 2-sided 95% confidence interval (CI) was calculated using the product limit method.
Time Frame: 1, 2 and 3 years after randomization
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 222
Percent probability
  1 year survival probability | 92.7 [89.8 to 94.7] | 94.9 [91.0 to 97.2]
  2 year survival probability | 78.4 [74.1 to 82.0] | 82.5 [76.6 to 87.0]
  3 year survival probability | 69.8 [65.1 to 73.9] | 65.0 [58.0 to 71.1]

16. Secondary Outcome: Number of Participants With Laboratory Abnormalities by Maximum Common Terminology Criteria for Adverse Events (CTCAE) Grade
Description: Laboratory abnormalities included anemia, hemoglobin increased, neutrophils (absolute), platelets, white blood cells, alanine aminotransferase (ALT), alkaline phosphatase, aspartate aminotransferase (AST), bilirubin (total), creatinine, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypokalemia, hypomagnesemia and hyponatremia. Laboratory abnormalities were graded by CTCAE version (v) 4.0 as Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = life-threatening. Categories with at least 1 non-zero data values are reported.
Time Frame: From randomization up to 28 days after last dose of study drug (assessed up to analysis date of 15-Nov-2021, approximately 8.7 years)
Population: AT population included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
Number analyzed (Participants) | 444 | 221
Participants
  Anemia: Grade 1-2 | 328 | 90
  Anemia: Grade 3 | 30 | 6
  Hemoglobin Increased: Grade 1-2 | 14 | 25
  Hemoglobin Increased: Grade 3 | 1 | 0
  Neutrophils (Absolute): Grade 1-2 | 109 | 42
  Neutrophils (Absolute): Grade 3 | 254 | 2
  Neutrophils (Absolute): Grade 4 | 60 | 1
  Platelets: Grade 1-2 | 289 | 32
  Platelets: Grade 3 | 6 | 0
  Platelets: Grade 4 | 1 | 0
  White Blood Cells: Grade 1-2 | 248 | 57
  White Blood Cells: Grade 3 | 177 | 0
  White Blood Cells: Grade 4 | 6 | 0
  ALT: Grade 1-2 | 222 | 76
  ALT: Grade 3 | 16 | 0
  ALT: Grade 4 | 1 | 0
  Alkaline Phosphatase: Grade 1-2 | 174 | 95
  Alkaline Phosphatase: Grade 3 | 7 | 0
  AST: Grade 1-2 | 260 | 82
  AST: Grade 3 | 23 | 2
  Bilirubin (Total): Grade 1-2 | 33 | 11
  Bilirubin (Total): Grade 3 | 3 | 0
  Creatinine: Grade 1-2 | 418 | 201
  Creatinine: Grade 3 | 8 | 0
  Creatinine: Grade 4 | 2 | 0
  Hypercalcemia: Grade 1-2 | 111 | 54
  Hypercalcemia: Grade 3 | 1 | 2
  Hyperkalemia: Grade 1-2 | 118 | 51
  Hyperkalemia: Grade 3 | 6 | 1
  Hyperkalemia: Grade 4 | 2 | 0
  Hypermagnesemia: Grade 1-2 | 71 | 26
  Hypermagnesemia: Grade 3 | 9 | 6
  Hypermagnesemia: Grade 4 | 2 | 0
  Hypernatremia: Grade 1-2 | 94 | 35
  Hypernatremia: Grade 3 | 8 | 1
  Hypoalbuminemia: Grade 1-2 | 118 | 42
  Hypoalbuminemia: Grade 3 | 2 | 0
  Hypocalcemia: Grade 1-2 | 158 | 48
  Hypocalcemia: Grade 3 | 4 | 1
  Hypocalcemia: Grade 4 | 3 | 0
  Hypokalemia: Grade 1-2 | 105 | 32
  Hypokalemia: Grade 3 | 11 | 2
  Hypomagnesemia: Grade 1-2 | 127 | 41
  Hypomagnesemia: Grade 3 | 1 | 0
  Hypomagnesemia: Grade 4 | 2 | 0
  Hyponatremia: Grade 1-2 | 107 | 44
  Hyponatremia: Grade 3 | 11 | 4

ADVERSE EVENTS:
Time Frame: From the date of randomization up to 28 days after last dose of study medication (final analysis till study completion, approximately up to 10.51 years)
Description: Same event may appear as non-SAE and SAE but are distinct events. Event may be an SAE in 1 participant and non-SAE in other, or participant may have both non-SAE and SAE. AT population included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received.
Arm/Group | Palbociclib Plus Letrozole | Placebo Plus Letrozole
All-Cause Mortality (participants affected / at risk) | 16/444 | 6/222
Serious Adverse Events (participants affected / at risk) | 125/444 | 38/222
Other Adverse Events (participants affected / at risk) | 435/444 | 209/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib Plus Letrozole (N=444) | Placebo Plus Letrozole (N=222)
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 3 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Dry age-related macular degeneration (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 2 | 0
Myopia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 1
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 4 | 0
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 1
Incarcerated hernia (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 3 | 1
Puncture site pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Serositis (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 5
Pyelonephritis (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 1 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Cataract traumatic (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bell's palsy (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 3 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Organic brain syndrome (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Stag horn calculus (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib Plus Letrozole (N=444) | Placebo Plus Letrozole (N=222)
Anaemia (Blood and lymphatic system disorders) | 125 | 23
Leukopenia (Blood and lymphatic system disorders) | 115 | 2
Neutropenia (Blood and lymphatic system disorders) | 308 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 64 | 4
Cataract (Eye disorders) | 28 | 7
Dry eye (Eye disorders) | 28 | 10
Lacrimation increased (Eye disorders) | 33 | 2
Vision blurred (Eye disorders) | 23 | 7
Abdominal distension (Gastrointestinal disorders) | 21 | 14
Abdominal pain (Gastrointestinal disorders) | 67 | 15
Abdominal pain upper (Gastrointestinal disorders) | 41 | 20
Constipation (Gastrointestinal disorders) | 105 | 36
Diarrhoea (Gastrointestinal disorders) | 136 | 51
Dry mouth (Gastrointestinal disorders) | 28 | 12
Dyspepsia (Gastrointestinal disorders) | 52 | 29
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 37 | 8
Nausea (Gastrointestinal disorders) | 169 | 59
Stomatitis (Gastrointestinal disorders) | 76 | 15
Toothache (Gastrointestinal disorders) | 23 | 7
Vomiting (Gastrointestinal disorders) | 80 | 37
Asthenia (General disorders) | 86 | 27
Chest pain (General disorders) | 31 | 7
Chills (General disorders) | 24 | 7
Fatigue (General disorders) | 183 | 65
Influenza like illness (General disorders) | 36 | 11
Mucosal inflammation (General disorders) | 49 | 9
Oedema peripheral (General disorders) | 65 | 19
Pain (General disorders) | 44 | 20
Pyrexia (General disorders) | 63 | 20
Bronchitis (Infections and infestations) | 27 | 7
Influenza (Infections and infestations) | 24 | 6
Nasopharyngitis (Infections and infestations) | 95 | 25
Oral herpes (Infections and infestations) | 31 | 3
Rhinitis (Infections and infestations) | 24 | 0
Sinusitis (Infections and infestations) | 30 | 9
Upper respiratory tract infection (Infections and infestations) | 75 | 26
Urinary tract infection (Infections and infestations) | 71 | 20
Contusion (Injury, poisoning and procedural complications) | 24 | 6
Fall (Injury, poisoning and procedural complications) | 60 | 18
Alanine aminotransferase increased (Investigations) | 65 | 13
Aspartate aminotransferase increased (Investigations) | 64 | 14
Blood creatinine increased (Investigations) | 33 | 8
Neutrophil count decreased (Investigations) | 106 | 7
Platelet count decreased (Investigations) | 38 | 1
Weight decreased (Investigations) | 30 | 10
White blood cell count decreased (Investigations) | 83 | 4
Decreased appetite (Metabolism and nutrition disorders) | 86 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 187 | 89
Back pain (Musculoskeletal and connective tissue disorders) | 117 | 52
Bone pain (Musculoskeletal and connective tissue disorders) | 45 | 24
Muscle spasms (Musculoskeletal and connective tissue disorders) | 46 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 37 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 65 | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 27 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 99 | 41
Dizziness (Nervous system disorders) | 80 | 34
Dysgeusia (Nervous system disorders) | 37 | 7
Headache (Nervous system disorders) | 109 | 62
Paraesthesia (Nervous system disorders) | 26 | 9
Anxiety (Psychiatric disorders) | 45 | 27
Depression (Psychiatric disorders) | 39 | 21
Insomnia (Psychiatric disorders) | 73 | 30
Breast pain (Reproductive system and breast disorders) | 24 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 127 | 48
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 80 | 35
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 43 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 50 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 150 | 36
Dry skin (Skin and subcutaneous tissue disorders) | 66 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 49 | 11
Rash (Skin and subcutaneous tissue disorders) | 79 | 24
Hot flush (Vascular disorders) | 101 | 69
Hypertension (Vascular disorders) | 45 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT01740427/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT01740427/SAP_001.pdf